CLINICAL TRIAL: NCT06339684
Title: HPV Immunological Markers of Cervical Persistent Infection and Oncogenesis
Acronym: HPVImmuno
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Daniele Lilleri, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: 2021 0075257
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-04

CONDITIONS: HPV-Related Cervical Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Whole blood and cervical samples (vaginal washing, cervical biopsy and pap-smear)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this observational study is to build an immunological assay to quantify an immunoscore system for clinical practice, which could identify HPV lesions with a risk of persistent cervical infection, which represents the main predictive factor of neoplastic evolution. A pattern of host immunological factors and HPV-related parameters, in order to identify an algorithm of risk stratification and tailoring treatment will be identified. Finally, in patients with HPV infection, a virus specific immunity after vaccination will be quantified, in order to highlight those patients who have the most significant risk of infection persistence.

DETAILED DESCRIPTION:
The end point of this study is to analyze host factors, including virus-specific immunity and HPV-related parameters influencing the onset and progression of squamous intraepithelial lesion (SIL), in order to define risk stratification and tailoring treatment, developing widely accessible and non-invasive assays immunoscore with high predictive value.

The progression of squamous intraepithelial lesion (H SIL) at 2 years in women with abnormal pap smear will also be evaluated (primary end point) and the immune host profile after anti-HPV prophylactic and therapeutic vaccination, in women with squamous intraepithelial lesions and with persistence of infection will be analyzed (secondary end point).

The investigators will analyze the patients, enrolled prospectively with abnormal pap smear every six months up to two years after diagnosis. At each time point, during colposcopy, peripheral blood (30 mL) and cervical samples (vaginal washing, cervical biopsy and pap-smear) will be collected for the characterization of local and peripheral immune response. Viral load, HPV integration will be assessed on cytological and tissue samples obtained from the patients at time of diagnosis and/or curative surgery.

For the secondary endpoints, the investigators will enroll patients with confirmed HPV infection, undergoing therapeutic and prophylactic HPV vaccination. The vaccination will be performed immediately after HPV lesion diagnosis. Follow-up program implies colposcopy every six months for 2 years. The investigators will analyze HPV-specific immune response every six months, and viral load and HPV integration at the time of diagnosis and at the end of the follow-up.

To evaluate antigen-specific proliferative response, PBMCs will be stimulated in triplicate in 96-well round-bottom plates with antigens L1, E6, E7 proteins of HPV- 16 and -18 and human Actin peptide pools for 7 days. Culture medium was RPMI 1640 supplemented with 2 mM L-glutamine, 100 U/mL penicillin and 100 µg/mL streptomycin solution, 10% of heat inactivated FBS, 1 mM Sodium Pyruvate, 100 µM non-essential amino acids, and 50 µM 2-Mercaptoethanol. After culture, cells will be washed, stained with Live/Dead Fixable Violet Dye ) and subsequently with CD3, CD4, CD8, CD25, CD278 (ICOS). Finally, cells will be washed and resuspended in PBS 1% paraformaldehyde.

A Cell Proliferation Index (CPI) for antigen-specific expanded T-cells will be determined by subtracting the percentage of CD25+ICOS+ CD3+CD4+ or CD3+CD8+ detected in PBMC incubated with actin peptides from the percentage of CD25+ICOS+ T-cell subsets detected in PBMC incubated with HPV peptides. A CPI <1.5% will be considered negative while a value ≥1.5% will be considered positive.

Flow cytometry analyses were performed with a FACS Canto II flow cytometer and BD DIVA software.

For the analysis of HPV-related features, molecular approaches will be used. HPV DNA will be extracted from biopsies and lesion swabs using automatized systems after specific lysis treatment for tissues.

HPV DNA will be then quantified using real time PCR specific for L1/E2 and E6 regions; in detail MY 09/11 fragment of L1 gene will be used. Results will be expressed as the number of copies/100.000 cells and normalized using a housekeeping gene.

For the differential quantification of integrated or episomal HPV DNA a specific standardized system for the amplification of ORF E2 and E6 will be used.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years.
* Abnormal PAP test
* HPV DNA positive

Exclusion Criteria:

* Inability to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be identified among women with abnormal PAP test undergoing colposcopy at Fondazione IRCCS Policlinico San Matteo.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2026-03-08 (Estimated); Study Completion 2026-03-08 (Estimated)

PRIMARY OUTCOMES:
Analysis plan for primary end-point | Time 0 (enrollment), Time 1 (6 months after colposcopy), Time 2 (12 months after colposcopy), Time 3 (18 months after colposcopy) and T4 (24 months after colposcopy)
  Univariable and multivariable interval-censoring Cox models will be applied to estimate the hazard ratios (HRs) of progression (advanced high grade lesions) at 2 years according to HPV-specific T cell response and HPV viral load measured at time of diagnosis. The best model will be selected based on Accuracy, Sensitivity, Specificity and Area Under Curve (AUC). LogRRs derived from the best model will be rounded to the closest integer and used to create a predictive score. Clustered sandwich estimator will be used to estimate standard errors, in order to account for the intra-patient correlation.

SECONDARY OUTCOMES:
Analysis plan for secondary end-points | Follow-up program implies colposcopy every six months for 2 years
  The effect of HPV Vaccine on progression will be analyzed by univariable and multivariable interval-censoring Cox models at six months after vaccination. Vaccine will be analyzed as a time dependent covariate. All analyses will be performed using the Stata software (release 16,StataCorp, College Station, TX, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gardella, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No